CLINICAL TRIAL: NCT01637740
Title: Pseudoexfoliation Syndrome in Myopes Defined With Optical Low Coherence Reflectometry
Brief Title: Pseudoexfoliation Syndrome in Myopes
Status: Completed | Type: Observational
Sponsor: General Hospital Sveti Duh (Other)
Responsible Party: Principal Investigator, Mladen Busic, M.D., PhD, General Hospital Sveti Duh
Other Study IDs: 04072012MB; 04072012UECUHSD (Other: University Eye Clinic, University Hospital "Sveti Duh")
Record Dates: First submitted 2012-07-07; First posted 2012-07-11 (Estimated); Last update posted 2012-07-11 (Estimated); Status verified 2012-07

CONDITIONS: Pseudoexfoliation Syndrome in Cataract Myopic Eyes
Keywords: myopia; pseudoexfoliation syndrome; optical low coherence reflectometry; ocular optical components; cataract
MeSH Terms: conditions — Myopia; Exfoliation Syndrome; Cataract

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective

GROUPS / COHORTS (2):
- eyes with pseudoexfoliation syndrome: cataract myopic eyes with pseudoexfoliation syndrome
- eyes without pseudoexfoliation syndrome: cataract myopic eyes without pseudoexfoliation syndrome

SUMMARY:
A retrospective study of 5753 eyes of cataract surgery patients was conducted at our Clinic. Ocular optical components measured by optical low coherence reflectometry biometer LENSTAR LS 900® of the cataract myopic eyes with pseudoexfoliation syndrome were put in comparison with those of cataract myopic eyes group without pseudoexfoliation syndrome.

DETAILED DESCRIPTION:
A retrospective study of 5753 eyes of cataract surgery patients was conducted at investigators Clinic in a period of 2.5 years. Pseudoexfoliation syndrome was found in 255 eyes. There were only 26 cataract myopic eyes with pseudoexfoliation syndrome. Refractive eye state was defined by preoperatively calculated emmetropization intraocular lens (IOL) value done by optical low coherence reflectometry biometer LENSTAR LS 900®. Ocular optical components of the cataract myopic eyes with pseudoexfoliation syndrome measured by this biometer were put in comparison with matched cataract myopic eyes group without pseudoexfoliation syndrome that have emmetropization IOL value within the same range as the cataract myopic eyes with pseudoexfoliation syndrome.

ELIGIBILITY:
Inclusion Criteria:

* cataract surgery patients ≥ 40 years old

Exclusion Criteria:

* cataract surgery patients < 40 years old

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 5753 eyes of cataract surgery patients ≥ 40 years old
Sampling Method: Probability Sample
Enrollment: 5753 (Actual)
Dates: Start 2009-08; Primary Completion 2012-01 (Actual); Study Completion 2012-01 (Actual)